CLINICAL TRIAL: NCT06887491
Title: The Effect of Dual-tasking Program on Cognitive and Physical Functions and Independence in Activities of Daily Living in Children With Duchenne Muscular Dystrophy: A Single-blind Randomized Controlled Trial
Acronym: DMD-DUAL-FUNC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Başak Çağla Arslan, Instructor, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 324S053; 324S053 (Other Grant/Funding Number: The Scientific and Technological Research Council of Türkiye)
Record Dates: First submitted 2025-03-09; First posted 2025-03-20 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: dual task; activity; cognitive; physical
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Individuals in the control group will be enrolled in a classical physiotherapy program.
  Interventions: Other: Conventional physiotherapy program
- Intervention (Experimental): Individuals in the intervention group will be enrolled in a dual task program in addition to the classical physiotherapy program.
  Interventions: Other: Conventional physiotherapy program + Dual task program

INTERVENTIONS:
Other: Conventional physiotherapy program — Breathing exercises such as thoracic extension Stretching exercises for upper and lower extremity muscles Active-assisted, active and low resistance exercises for lower and upper extremity muscles according to muscle strength They will be asked to perform a home program including functional exercises (going up and down stairs, taking steps, etc.) at least 5 days a week, 2 times a day. The exercises will be checked by phone once a week and regular participation in the program will be ensured.
  Arms: Control
Other: Conventional physiotherapy program + Dual task program — Breathing exercises such as thoracic extension Stretching exercises for upper and lower extremity muscles Active-assisted, active and low resistance exercises for lower and upper extremity muscles according to muscle strength They will be asked to perform a home program including functional exercises (going up and down stairs, taking steps, etc.) at least 5 days a week, 2 times a day. The exercises will be checked by phone once a week and regular participation in the program will be ensured.
  Dual task program: Walking 10 meters (Single task) and basic dual task introduction. Simple motor-motor tasks (e.g., holding a ball while walking). Carrying a half-full water bottle in each hand while walking. Placing or carrying objects accompanied by exercises requiring balance. Counting Counting backwards while walking. Solving simple math problems while walking Complexification of motor-motor and cognitive-motor tasks.
  Dual tasks similar to activities of daily living
  Arms: Intervention

SUMMARY:
Duchenne Muscular Dystrophy (DMD) is an X-linked recessive disorder characterized by progressive muscle degeneration and frequent developmental, cognitive and behavioral impairments, occurring in one in 5000 live births of boys. DMD is caused by a deficiency of the protein dystrophin, which maintains the structure and functionality of muscle cells. The absence of dystrophin leads to the weakening and eventual death of muscle cells, resulting in reduced muscle strength and impaired motor function. In early childhood, children with DMD may experience delays in basic motor skills such as walking and standing. Later in life, the disease leads to more severe motor dysfunctions, including loss of muscle strength, problems with balance and coordination, and an increased risk of falls.

DMD can also negatively affect cognitive function. Dystrophin is found not only in muscles but also in the brain, and its deficiency in the brain can lead to cognitive problems such as learning disabilities, attention deficits and impaired executive function. These cognitive impairments can affect the academic performance of children with DMD and their functional abilities in everyday life.

In this project, the potential effects of a dual task program designed for children with DMD on physical and cognitive functioning will be examined. Dual task training aims to increase children's capacity to perform two different tasks simultaneously, which may improve the integration of cognitive and motor functions. For example, activities such as counting while walking or answering a question while carrying an object in the hand require children to use both motor and cognitive skills simultaneously. Such exercises can increase coordination between cognitive and motor functions and improve the independence of children with DMD in activities of daily living and their overall quality of life.

The main goals of the program are to produce positive effects on motor skills and cognitive functions, improve balance and coordination, and enable children to move more independently in activities of daily living. Furthermore, this study highlights the value of a multidisciplinary approach, providing important insights into how rehabilitation approaches can be developed for individuals with a special condition such as DMD. Collaboration between physiotherapists and occupational therapists plays a critical role in providing comprehensive care for these children.

The methodology of this study included boys with DMD who were admitted to Lokman Hekim University Muscular and Nerve Diseases Application Center. The children will be randomly assigned to the intervention and control groups, and the children in the intervention group will be enrolled in a dual task performance program for two days a week, one session a day, 45 minutes each session, for eight weeks, with at least two days in between. The effectiveness of the program will be measured using various motor and cognitive assessment tools.

The hypotheses of this study are that dual task training will positively affect motor and cognitive and physical functions in children with DMD, improve balance and coordination, and increase the level of independence of these children in activities of daily living. In conclusion, this project aims to contribute to the development of innovative approaches in the treatment of children with DMD. This approach can improve the overall quality of life of children, as well as support their social participation and educational achievement.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is an X-linked recessive disorder characterized by progressive muscle degeneration, as well as frequent developmental, cognitive, and behavioral impairments, with a prevalence of one in 5,000 live male births. It is caused by mutations in the dystrophin gene, leading to the absence or severe deficiency of dystrophin, a cytoskeletal protein essential for the strength, stability, and functionality of myofibrils. Although boys with DMD appear normal at birth, difficulties in developmental milestones such as independent walking and standing become apparent during early childhood. Around the age of four, proximal muscle weakness, particularly in the hips, becomes evident due to the progressive damage to skeletal muscles resulting from dystrophin deficiency, often manifesting as Gower's sign. As the disease advances, postural and balance impairments, reduced endurance, and deficiencies in functional skills emerge. The progressive decline in muscle strength and endurance further diminishes physical activity capacity while increasing the energy expenditure required for activities, resulting in a higher frequency of falls. Despite improvements in the survival rates of individuals with DMD, the progression of the disease is inevitable and typically leads to the loss of ambulation and the need for a wheelchair by ages 11 to 12, accompanied by significant physical dependence.

DMD affects not only neuromuscular but also cognitive functions, a phenomenon first observationally described by Duchenne de Boulogne in 1868 and subsequently corroborated by numerous studies. High levels of dystrophin are found in nerve cells of the cerebral cortex, cerebellum, and hippocampus, regions critical for learning and memory functions. Mutations impacting distal regions, such as Dp140 and Dp71, are associated with lower IQ levels, while proximal mutations contribute to cognitive challenges. The anatomical areas affected by these mutations are connected to the frontal lobe, which is responsible for executive functions such as memory, future planning, decision-making, reasoning, and sustained attention. Magnetic resonance imaging studies have revealed that the lack of dystrophin impacts not only muscles but also the brain, with cognitive impairments observed in approximately one-third of boys with DMD. These impairments are non-progressive and include a mean IQ approximately one standard deviation below the norm. Verbal intelligence quotient scores are often more affected than performance scores. Common cognitive features in DMD include deficits in attention components, short-term verbal memory (working memory), executive functions, expressive language, reading skills, and delays in language acquisition. Nearly half of individuals with DMD experience learning difficulties, and conditions such as borderline intellectual functioning, autism spectrum disorders, attention deficit hyperactivity disorder (ADHD), epilepsy, and anxiety occur more frequently compared to the general pediatric population.

Dual-tasking refers to the simultaneous execution of two tasks that can also be performed independently, each serving a distinct purpose. Examples include walking while talking, carrying a bag while walking, or thinking about items on a shopping list while navigating a store. The capacity to perform such dual tasks, known as dual-task performance, is integral to participation in daily life. Dividing attention between two concurrent tasks often leads to a decrease in performance in one or both tasks compared to performing them individually, a phenomenon referred to as dual-task interference. Factors such as task difficulty and the allocation of attention disproportionately to one task influence dual-task interference. Dual-task performance can be categorized into motor-motor, cognitive-cognitive, and cognitive-motor tasks.

Although dual-tasking has been extensively studied in adults, research on pediatric populations remains limited. Studies involving children often assess parameters such as walking speed, cadence, stride length, double-support time, and step width during tasks like walking while counting. Compared to adults, children experience greater dual-task interference, attributed to the ongoing development of the central nervous system, which governs motor and cognitive processes. In modern daily life, children increasingly engage in dual-tasking, combining activities such as eating, doing homework, or performing household chores with watching television, playing video games, or texting. Studies investigating dual-task performance in children with DMD have reported that impairments in functional status and balance control adversely affect their dual-task capabilities. Cognitive challenges such as attention, short-term memory, and executive function deficiencies exacerbate performance issues in one or both tasks during dual-tasking. Additionally, cognitive-motor dual tasks have a significant impact on functional mobility scores in children with DMD compared to their typically developing peers. Incorporating dual-task evaluations into rehabilitation processes is crucial for guiding management strategies and improving outcomes.

Research exploring the effects of dual-task programs on cognitive, motor, and physical functions in children demonstrates promising results for enhancing various developmental domains. Studies in children with spastic diplegia, intellectual disabilities, and cerebral palsy, as well as those recovering from traumatic brain injuries, highlight improvements in balance, gross motor functions, and functional mobility following dual-task training programs. These findings underscore the potential therapeutic value of dual-task programs for fostering development and functional outcomes in children with various conditions. However, no studies to date have specifically examined the cognitive and physical effects of dual-task programs in children with DMD. Therefore, this project aims to investigate the impact of a dual-task program on the cognitive and physical functions, as well as the independence in daily living activities, of children with DMD.

Aim of the Project The primary aim of this project is to determine the potential benefits of a dual-task program on the cognitive and physical functions of children diagnosed with Duchenne Muscular Dystrophy (DMD) and to explore how such training can be integrated into rehabilitation programs. Additionally, the project seeks to investigate how this approach affects the performance, independence, and quality of life of children in daily living activities.

Objectives of the Project Improvement of Motor and Cognitive Functions: It is anticipated that dual-task training will have positive effects on the motor skills and cognitive functions of children. Specifically, dual-task training may support the more effective use of motor skills by enhancing cognitive functions such as attention and memory.

Enhancement of Balance and Coordination: Dual-task training has the potential to improve children's balance and coordination, resulting in reduced fall risk and better overall physical performance during daily living activities.

Increase in Independence Levels: Following training, improvements in the ability of children to move more independently in daily life activities are expected, contributing to an enhanced quality of life.

Significance of the Project Understanding the impact of such a program on individuals with a specific condition like DMD is critical for optimizing rehabilitation approaches. The findings may lead to the development of more effective treatment plans tailored to the progression of the disease and the specific needs of the individual. With advancements in technology and rehabilitation practices, the expected increase in life expectancy of individuals with DMD, alongside a rise in situations requiring cognitive function, underscores the growing importance of cognitive rehabilitation. This approach is also relevant in addressing future challenges in employment and career development.

Dual-task training is particularly significant for physiotherapists and occupational therapists. Through these programs, individuals can develop the ability to perform two tasks simultaneously. Physiotherapists can utilize dual-task programs to reduce fall risks and enhance multitasking abilities, particularly in neurological and geriatric patients during walking, balance, and neurological rehabilitation. Occupational therapists, on the other hand, help individuals perform daily living activities more efficiently by strengthening cognitive functions and improving adaptation skills. In both professions, the shared goal of dual-task programs is to enhance patients' independence and quality of life, reduce fall risks, and improve both cognitive and motor functions. This program equips patients to better manage the challenges encountered in daily life. Consequently, this study is valuable for occupational therapists and physiotherapists as it emphasizes the importance of a multidisciplinary approach, promotes innovative methods in professional practice, and has the potential to advance rehabilitation strategies for individuals with specific conditions like DMD.

Contributions to Current Rehabilitation Practices The rehabilitation of children with DMD typically involves approaches such as physiotherapy, muscle strengthening, respiratory exercises, and stretching, which are often single-task focused. However, these approaches do not sufficiently address the dual-task scenarios frequently encountered in daily life.

Dual-task programs aim to enhance the ability to perform combined cognitive-motor tasks often required in daily living. This approach seeks to improve children's independence, balance, motor skills, and cognitive functions in everyday activities. Moreover, due to the progressive nature of DMD, children may avoid dual-task scenarios over time, potentially leading to increased inactivity. By addressing this, dual-task training can help overcome kinesiophobia and reduce fear of movement.

The findings of this project can be integrated into clinical practice, recommending the inclusion of dual-task programs in rehabilitation protocols. This integration has the potential to improve the overall quality of life of children with DMD and support their long-term independence.

ELIGIBILITY:
Inclusion Criteria:

* Being a boy between the ages of 6-12 years who has been diagnosed with DMD as a result of specialist evaluation and gene analysis,
* Being in stage 1 and stage 2 according to Vignos lower extremity classification,
* A score of 27 and above on the Modified Mini-Mental Test,
* To have the ability to walk at least 10 meters independently,
* Receiving at least 8 physiotherapy and rehabilitation sessions for 1 month,
* Volunteering to participate in the study by their parents and reading and signing the informed consent form.

Exclusion Criteria:

* Having a neurological disease other than DMD and/or another diagnosed neurological disease accompanying DMD,
* To have had any injury and/or surgery within the last six months,
* Having a co-operation problem that prevents completing the assessments for any reason,
* Having difficulty understanding and speaking the Turkish language.

Ages: 6 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-16 (Estimated)

PRIMARY OUTCOMES:
Demographic information form | Baseline
  Age (years), height (centimeters), body weight (kilograms) and body mass index (BMI) values of the children will be recorded. From the families of children with DMD, a detailed history of the disease will be obtained, including medical history, surname, DNA analysis result, age at diagnosis (years) and steroid use (name of steroid, dose, year of use), presence of scoliosis (if any, degree, year of onset) and functional status of the patient.
Modified Mini-Mental Test | Baseline
  The Modified Mini-Mental State Test (MMSE) will be used to evaluate the cognitive levels of children. Originally designed to identify cognitive impairments in adults, it is a quick and reliable tool with Turkish validity. While numerous neuropsychological tests are available for assessing cognitive skills in children, their lengthy administration and the need for professional expertise often limit their usability. The MMSE was therefore adapted with minor modifications for pediatric use and has been applied in children with DMD. This version assesses attention, orientation, memory, language skills, the ability to follow verbal and written commands, reading and writing abilities, and copying drawings. The test is scored out of 37, with values below 27 indicating potential mental retardation or dementia. Its simplicity and efficiency make it a practical choice for screening cognitive functions in children.
Dual task assessment | Baseline and 2 months
  In the intervention group, dual-task performance will be evaluated in the first and last sessions, while the control group will be assessed eight weeks apart. The study includes motor-motor and cognitive-motor tasks, commonly used combinations in dual-task evaluations. The primary task is a 10-meter walk. The motor-motor task involves walking while carrying two 500 ml half-full bottles, considering the muscle weakness in children with DMD. The cognitive-motor tasks include backward counting, adapted to the child's age (e.g., a 6-year-old counts backward by ones from 10, a 12-year-old by sevens from 100) and recalling five previously provided age-appropriate words during the walk. The order of word recall is unimportant; any words remembered are recorded, and missed words are noted. Dual-task effect (DTE) will be calculated using the formula:
  DTE = ((dual-task performance - single-task performance) / single-task performance) × 100 Children will equally prioritize both tasks. Measuremen
Dynamic Occupational Therapy Cognitive Assessment-Child Version (DOTCA-ch) | Baseline and 2 months
  Developed by occupational therapists in 2004 as "Dynamic Occupational Therapy Cognitive Assessment-Child (DOTCA-ch)", the test was designed to assess the cognitive abilities and learning potential of children aged 6-12 years. As a performance-based test, the DOTCA-Ch has a different style in which children actively perform their cognitive assessments and, when deemed appropriate, can perform the test with help, and is frequently preferred by therapists. The assessment domains of the ADAS-C are processing speed, comprehension/problem solving, apraxia, attention/working memory, cognition and executive functions. It consists of 22 subtests in five cognitive domains (orientation, spatial perception, praxis, visual-motor interpretation and thinking processes). Five of the subtests of the Visual-Motor Interpretation test test test immediate and delayed memory.
Jebsen Taylor Hand Function Test | Baseline and 2 months
  In this test, a total of 7 different activities are applied, including checkers, collecting 6 small objects, feeding simulation, card spinning, carrying empty jars, carrying full jars and writing activities. The person will be asked to perform these activities with the dominant upper limb and the assessor will record the completion times of the activities.
6 Minute Walk Test | Baseline and 2 months
  The 6-minute walk test (6MWD), which has proven validity and reliability in children with DMD, will be used to assess submaximal walking function and physical capacity. The distance the child walks for six minutes on a track with 25 meters between the start and end points will be recorded in meters. One researcher will walk with the child and ensure that the course is completed. Another researcher will record with a stopwatch, paper and pen to check the duration of each round and the total time. The 6DYT is a simple test to administer and is recognized as an important outcome measure for children with DMD
The Pediatric Berg Balance Scale | Baseline and 2 months
  The Pediatric Berg Balance Scale (PBBS) will be used to assess the balance of children. The PBBS is a 14-part test that includes parameters such as sitting to standing, standing, transfers, stepping, and turning and evaluates balance functionally. Each section is scored between 0-4 and the highest score that can be obtained from the scale is 56. High scores indicate good balance performance.
Pediatric Functional Independence Measure (WeeFIM) | Baseline and 2 months
  Pediatric Functional Independence Measure (WeeFIM) will be used to determine the independence level of children. WeeFIM consists of six sections and 18 items including self-care, sphincter control, transfers, locomotion, communication, social and cognitive domains, which are activities of daily living in children, and is administered by direct observation or interview with someone who can provide information about the child's performance. Each item is scored from complete independence (7 points) to fully assisted (1 point), with a minimum score of 18 (fully dependent) and a maximum score of 126 (fully independent). It is a quick and reliable scale suitable for use in the pediatric population, including children with DMD.
ACTIVLIM | Baseline and 2 months
  ACTIVLIM will be used to determine activity limitations in children with DMD. ACTIVLIM is a scale that can be used in all age groups to assess activity limitations in neuromuscular diseases and has Turkish validity and reliability. There are 22 items in total in the scale that evaluates activities of daily living that require the use of upper and lower extremities. In the scoring of the scale, 0= cannot do the activity, 1= has difficulty in doing the activity, 2= can do the activity easily and higher scores indicate less activity limitation.
The Pediatric Quality of Life Inventory (PedsQLTM) 3.0 Neuromuscular module | From enrollment to the end of treatment at 8 weeks
  The Turkish version of the Pediatric Quality of Life Inventory (PedsQLTM) 3.0 Neuromuscular module will be used to assess the quality of life of children with DMD. The PedsQLTM 3.0 Neuromuscular Module was created to assess quality of life in neuromuscular disorders such as DMD and SMA. The module consists of 25 items and has 3 subcategories: About My Neuromuscular Disease (17 items), Communication (3 items), About Family Resources (5 items). The PedsQLTM assesses the health-related quality of life of children with chronic diseases from the perspective of both the child and the family. The PedsQL scale, which is a questionnaire designed for children aged 2-18 years, has specialized forms for 2-4, 5-7, 8-12, 13-18 age ranges. Considering the inclusion criteria, the PedsQL scales developed for the 5-7 and 8-12 age ranges will be used in our study
Pediatric Quality of Life Inventory (PedsQL)- Multidimensional Fatigue Scale | From enrollment to the end of treatment at 8 week
  Pediatric Quality of Life Inventory (PedsQL)- Multidimensional Fatigue Scale will be used to assess the fatigue levels of children with DMD. The PedsQL-Multidimensional Fatigue Scale consists of 3 subsections and 18 items: General Fatigue (6 items), Fatigue during Sleep/Rest (6 items) and Cognitive Fatigue (6 items). The scale is scored on a 5-point Likert scale: Never: 0, Almost never: 1, Sometimes: 2, Frequently: 3, Always: 4. As a score, it is scored as 0=100, 1=75, 2=50, 3=25, 4=0 in the hundred point system. While a score can be calculated separately for each subsection, the total score is obtained by summing the scores obtained from the sections. High scores indicate low fatigue. The PedsQL-Multidimensional Fatigue Scale has child and parent forms for 2-4 years, 5-7 years, 8-12 years, and 13-18 years separated according to different age groups. In our study, the 5-7 and 8-12 years old child and parent form will be used to eval

OTHER OUTCOMES:
Vignos lower extremity classification | Baseline
  The functional level of the lower extremities of children with DMD will be evaluated with the "Vignos lower extremity classification". Vignos lower extremity classification is a scale consisting of 10 stages developed to evaluate the ambulation level in neuromuscular diseases. In this scale, the ambulation level of the person decreases as one moves from the first stage to the 10th stage. The staging of the Vignos lower extremity classification is as follows:
  Stage 1: Walks and climbs stairs without assistance. Stage 2: Walks and climbs stairs in less than 12 seconds by holding on to the handrail.
  Stage 3: Walks and climbs stairs slowly, holding on to the handrail, in more than 12 seconds.
  Stage 4: Can walk unassisted and get up from a chair, but cannot climb stairs. Stage 5: Can walk unassisted and get up from a chair, but cannot climb s
Brooke upper limb functional classification | Baseline
  The "Brooke upper extremity functional classification" used in neuromuscular diseases will be used to assess the functional level of the upper extremity. This classification is a staging system developed by Brooke et al. The classification consists of six stages and progression from the first stage to the sixth stage indicates a decrease in the functionality of the upper extremity. The stages of the Brooke Upper Extremity Functional Classification are as follows:
  Stage 1: Starts movement with the arms at the side and can fully join the hands above the head.
  Stage 2: However, he/she can bring his/her arms above his/her head by flexing his/her elbows or use auxiliary muscles.
  Stage 3: Cannot raise the hands above the head, but can bring the cup to the mouth (using both hands if necessary).
  Stage 4: Can raise hands to mouth, but cannot bring a glass of water to mouth. Stage 5: Cannot raise hand

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Cankaya, Turkey (Türkiye)